CLINICAL TRIAL: NCT02558335
Title: Circulating Tumor Markers for High Grade Glioma
Brief Title: CTCs for High Grade Glioma
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 09313
Record Dates: First submitted 2015-08-19; First posted 2015-09-24 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Stage III and IV Glioma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 22 cc of blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify and quantify circulating tumor markers, which are associated with the presence of tumors. The current imaging available does not allow specificity of tumor size as it relates to pseudoprogression (a temporary enlargement or "swelling" of the tumor after treatment before it shrinks). Our hope is that CTCs will provide a more accurate description of tumor state for high grade glioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven high grade glioma who are undergoing definitive radiotherapy as a part of their treatment regimen or patients with radiographic appearance of high grade glioma
* Age 18 or older
* Signed informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with grade III and IV glioma
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
to identify and quantify circulating tumor markers | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lustig, MD, Principal Investigator — Abramsvaniaon Cancer Center of the University of Pennsyl
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States